CLINICAL TRIAL: NCT04785040
Title: The Turkish Version of the Musculoskeletal Pain Intensity and Interference Questionnaire for Musicians (MPIIQM-T): A Validity, Reliability and Cross-cultural Adaptation Study
Brief Title: The Turkish Version of the Musculoskeletal Pain Intensity and Interference Questionnaire for Musicians (MPIIQM-T)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ankara Yildirim Beyazıt University (Other)
Responsible Party: Sponsor
Other Study IDs: 16.04.2021-44
Record Dates: First submitted 2021-03-03; First posted 2021-03-05 (Actual); Last update posted 2021-05-19 (Actual); Status verified 2021-05

CONDITIONS: Musculoskeletal Pain; Questionnaire
Keywords: musician; orchestra musicians; Musculoskeletal Pain; questionnaire
MeSH Terms: conditions — Musculoskeletal Pain

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 5 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1
  Interventions: Other: The groups evaluated by The Musculoskeletal Pain Intensity and Interference Questionnaire for Professional Orchestra Musicians, Brief Pain Inventory, QuickDASH and Fatigue Severity Scale

INTERVENTIONS:
Other: The groups evaluated by The Musculoskeletal Pain Intensity and Interference Questionnaire for Professional Orchestra Musicians, Brief Pain Inventory, QuickDASH and Fatigue Severity Scale — The groups evaluated by The Musculoskeletal Pain Intensity and Interference Questionnaire for Professional Orchestra Musicians, Brief Pain Inventory, QuickDASH and Fatigue Severity Scale

SUMMARY:
The aim of this study, original named "The musculoskeletal pain intensity and interference questionnaire (MPIIQM)" is the Turkish validation, reliability and cross-cultural validation of the questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* permanent musician in an orchestra
* understand and reading Turkish

Exclusion Criteria:

* freelance musician

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: professional orchestra musician
Sampling Method: Non-Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2021-04-16 (Actual); Primary Completion 2021-07 (Estimated); Study Completion 2021-07 (Estimated)

PRIMARY OUTCOMES:
The Musculoskeletal Pain Intensity and Interference Questionnaire for Professional Orchestra Musicians | Baseline
  The Musculoskeletal Pain Intensity and Interference Questionnaire for Professional Orchestra Musicians (MPIIQM) is a self-report questionnaire comprised of 22 items about performance-related musculoskeletal disorders (PRMD) in musicians. Age, gender and practice habits, different prevalence periods of PRMD, pain localization, pain intensity, pain interference are evaluated. The scoring of questionnaire is focused on the pain intensity and pain interference subscale. The pain intensity score can be defined as the sum of the four pain intensity items (0-40) or the mean of pain intensity score (0-10). The pain interference score can be defined as the sum of the five pain interference items (0-50) or the mean of pain interference score (0-10).
The Musculoskeletal Pain Intensity and Interference Questionnaire for Professional Orchestra Musicians | 5 days after
  The Musculoskeletal Pain Intensity and Interference Questionnaire for Professional Orchestra Musicians (MPIIQM) is a self-report questionnaire comprised of 22 items about performance-related musculoskeletal disorders (PRMD) in musicians. Age, gender and practice habits, different prevalence periods of PRMD, pain localization, pain intensity, pain interference are evaluated. The scoring of questionnaire is focused on the pain intensity and pain interference subscale. The pain intensity score can be defined as the sum of the four pain intensity items (0-40) or the mean of pain intensity score (0-10). The pain interference score can be defined as the sum of the five pain interference items (0-50) or the mean of pain interference score (0-10).

SECONDARY OUTCOMES:
Brief Pain Inventory | Baseline
  In Brief Pain Inventory, patients rate their pain severity and pain interference dimensions on a numeric rating scale from 0 to 10. In the inventory, a score of 1-4 is defined as mild pain, a score of 5-6 as moderate pain, and a score of 7-10 as severe pain.
The QuickDASH | Baseline
  The QuickDASH (Quick-Disabilities of the Arm, Shoulder and Hand Score) is a shortened version of the DASH (Disabilities of the Arm, Shoulder and Hand Score), featuring 11 instead of 30 items about physical function and symptoms in patients with musculoskeletal disorders of the upper extremities. 0-100 from each part of the Quick-DASH questionnaire (0 = no disability, 100 = most severe disability) is scored.
The Fatigue Severity Scale | Baseline
  The Fatigue Severity Scale (FSS) assess fatigue severity in a variety of medical conditions. It consists of 9 items rated on a 7-point Likert scale (1=strong disagreement, 7=strong agreement). High scores indicate fatigue. 28 points and above indicate the presence of severe fatigue.

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Yildirim Beyazit University, Ankara, Turkey (Türkiye)